CLINICAL TRIAL: NCT07145801
Title: Contrast-Enhanced Ultrasound Evaluation of Radioembolization Treatment Response
Brief Title: Y-90 Treatment Response Using Transarterial Radioembolization
Acronym: TARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, john eisenbrey, Principal Investigator, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0539; JT 45493 (Other: JeffTrial Number); 1R21CA303648 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: HCC; Hepatocellular Carcinoma; Liver Cancer; Hepatic Neoplasm; Primary Liver Cancer; Liver Neoplasm
Keywords: transarterial radioembolization; TARE; CEUS; contrast-enhanced ultrasound; hepatocellular; carcinoma; HCC; hepatocellular carcinoma (HCC); liver cancer; liver tumors; liver lesions; microbubbles; liver parenchyma; liver imaging; HCC locoregional therapy; Ultrasound; Kupffer; Yttrium-90; tumor viability; time intensity curves; parametric maps; microbubble destruction; bolus contrast injection; CEUS biomarker; Y90 TARE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CEUS with Lumason and Sonazoid (Experimental): The plan is to enroll a total of 30 patients scheduled for TARE of a treatment naïve HCC over an 18-month period, allowing for a minimum of 6 months follow up. Patients will undergo a CEUS examination within two weeks of their first two clinically indicated CT/MRI exams (obtained at Jefferson 1-2 months and 4-6 months post TARE).
  Interventions: Diagnostic Test: Lumason; Diagnostic Test: Sonazoid

INTERVENTIONS:
Diagnostic Test: Lumason — Following baseline ultrasound imaging, CEUS will be performed using dual B-mode and CEUS mode. For the first injection using Lumason the approximate tumor mid-line will be imaged during breath hold until complete tumor enhancement is achieved followed by imaging sweeps through the tumor. Intermittent imaging will be performed after that. Following a 10 minute Lumason wash-out period, participants will then receive a bolus injection of Sonazoid with identical imaging protocol to Lumason for the first 60 seconds to evaluate arterial phase enhancement. Imaging sweeps of the tumor will then be obtained at 1 and 2 minutes to evaluate enhancement within the late vascular phase to detect early washout. After visualization in the late phase, imaging will resume to evaluate the Kupffer phase of contrast enhancement. Following completion of the exam, patients will be monitored for at least 30 minutes before being discharged and all data will be exported for later off-line analysis
  Other Names: sulfur hexafluoride lipid-type A microspheres; SonoVue; SF6 lipid microspheres; Sulfur hexafluoride lipid microspheres; Sulfur Hexafluoride; SF₆ microspheres
Diagnostic Test: Sonazoid — Participants will receive a bolus injection up to (0.12 µl of MB/kg) of Sonazoid, followed by 5-10 ml of normal saline. Imaging of Sonazoid will be identical to the protocol described above for the first 60 seconds to evaluate arterial phase enhancement. Imaging sweeps (5-10 seconds) of the tumor will then be obtained in at 1 and 2 minutes to evaluate enhancement within the late vascular phase and detect early washout. After that imaging will resume to evaluate the Kupffer phase of contrast enhancement. Kupffer phase imaging (also called the postvascular phase) starts approximately 8-10 mins after injection when the free circulating microbubbles have been eliminated from the vasculature with Kupfer-cell enhancement persisting for up to 2 hours. Sonazoid CEUS will be performed in all patients after Lumason clearance from the circulation, usually within 15 min after injection.
  Other Names: Perflubutane; Perfluorobutane microbubbles; NC100100 acoustic contrast agent

SUMMARY:
This prospective clinical study will examine the ability of contrast-enhanced ultrasound (CEUS) to assess the treatment response of hepatocellular carcinoma (HCC) to transarterial radioembolization (TARE). HCC is the third leading cause of cancer mortality worldwide and the single fastest growing cause of cancer mortality in the United States. TARE is recommended for 15-25% of HCC patients. Treatment response is generally evaluated using contrast-enhanced Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) 1-2 months and 4-6 months post-TARE. Although TARE is an effective therapy, assessment of treatment response using CT/MRI is challenging because CT/MRI frequently diagnoses tumor response as equivocal or non-progressing for up to 6 months post-TARE based on Liver Imaging Reporting and Data System (LI-RADS) criteria. This delay in diagnosing tumor viability subsequently delays needed retreatment and can even serve as a barrier to transplantation. Our prior work in HCC locoregional therapy has shown CEUS provides improved sensitivity in detecting viable tumor following transarterial chemoembolization relative to traditional CT/MRI. Therefore, the investigators propose to evaluate both qualitative and quantitative CEUS as a tool for evaluating HCC post-TARE at similar time points of clinically recommended cross-sectional imaging, while also investigating the role of Kupffer phase imaging.

The investigator plans to enroll a total of 30 patients scheduled for TARE of a treatment naïve HCC over an 18-month period, allowing for a minimum of 6 months follow up. Patients will undergo a CEUS examination within two weeks of their first two clinically indicated CT/MRI exams (obtained at Jefferson 1-2 months and 4-6 months post TARE). Patients will be recruited across six major hospitals within the Jefferson Health Enterprise. Those eligible for participation will be identified by project co-investigators and contacted by the study coordinator to discuss participation and to explain the study. The patient will be given time to consider the risks and benefits of the study and ask questions about participation. If agreeable, the patient will then arrange with the project coordinator to come to Jefferson's center city campus to sign consent and take part in the research study.

DETAILED DESCRIPTION:
Following baseline ultrasound imaging, CEUS will be performed using dual B-mode and CEUS mode. For the first injection using Lumason the approximate tumor mid-line will be imaged during breath hold until complete tumor enhancement is achieved followed by imaging sweeps through the tumor. Intermittent imaging will be performed after that. Following a 10 minute Lumason wash-out period, participants will then receive a bolus injection of Sonazoid with identical imaging protocol to Lumason for the first 60 seconds to evaluate arterial phase enhancement. Imaging sweeps of the tumor will then be obtained at 1 and 2 minutes to evaluate enhancement within the late vascular phase to detect early washout. After visualization in the late phase, imaging will resume to evaluate the Kupffer phase of contrast enhancement. Following completion of the exam, patients will be monitored for at least 30 minutes before being discharged and all data will be exported for later off-line analysis.

A total of 30 patients scheduled for TARE of a treatment naïve HCC will be enrolled over an 18-month period, allowing for a minimum of 6 months follow up. Given our estimated volume of roughly 35 eligible patients per year, this provides a relative recruitment rate of 53% which is consistent with our prior studies in HCC [9,11]. Eligible patients will be screened from our intuition's multi-disciplinary HCC tumor board (led by co-I Dr. Civan with input from other co-I's Drs. Lyshchik, Topper, and Anton).

Eligible patients will be identified by the project coordinator (Ms. Bradigan, RN) using our electronic medical records system. Additionally, eligible patients will be identified by co-Investigators Dr. Anton (who heads our HCC locoregional treatment program), Dr. Topper (who also has a robust HCC locoregional therapy census), and Dr. Civan (who oversees the Jefferson liver tumor board and transplant program). Additionally, the NCT listing will be posted on the websites of Jefferson's Kimmel Cancer Center. Eligible patients will be asked to contact the study coordinator to discuss participation. Whenever possible, the attending physician will approach the patient to discuss interest in the study. The study research coordinator will then contact the patient to explain the study. The patient will be given time to consider the risks and benefits of the study and ask questions about participation. If agreeable, the patient will then arrange with the project coordinator to come to Jefferson's center city campus to sign consent and take part in the research study.

The subject population for this study will be made up of approximately 33% women based on the patient populations at our university scheduled for TARE. The patient population of this project will reflect the population demographics found at major American urban academic health centers. The overall demographics include 66% Caucasian, 30% African American, and 4% Asian, with 10% representing Hispanic patients. Stratified analyses will be performed of this clinical study to allow us to determine if there are clinically important sex/gender and/or race/ethnicity differences and allow us to target the optimal imaging strategy to a precisely defined patient population based upon patient demographics.

Importantly, this clinical study does not meet the NIH criteria for a clinical trial because the study is not designed to evaluate the effect of the intervention on the participants (i.e., clinical intervention will not be changed based on CEUS findings at this point).

Following informed consent, a full history and physical examination will be obtained from the patient's referring physician notes. Factors that might negatively affect diagnostic performance of CEUS (prior tumor size, depth, and anatomic location; presence of ascites; and body mass index) will be recorded for each patient. Participants will first undergo baseline ultrasound imaging. B-mode measurements and sweeps of the lesion in the transverse and sagittal planes will be acquired. Following B-mode imaging, power Doppler cine loops and volumes of the lesion of interest will be recorded in order to obtain unenhanced flow information.

Patients will undergo a CEUS examination within two weeks of their first two clinically indicated CT/MRI exams (obtained at Jefferson 1-2 months and 4-6 months post TARE). Ultrasound scanning will be performed by an accredited sonographer with >5 years of CEUS experience (Ms. Wessner) using a Logiq E10 scanner with C1-6 probe. When available, ultrasound-MR fusion may be used. CEUS imaging (first bolus contrast injection) will be performed using dual B-mode (used to locate anatomical features) and CEUS mode. A low mechanical index (MI < 0.13) will be used to minimize microbubble destruction during imaging. The standard nonlinear imaging frequency pairings in the CEUS software will be used (transmitting at 2 MHz and receiving at 4 MHz) and gain settings will be adjusted to minimize nonlinear signals prior to contrast injection. For Lumason (1.5-2.4 ml bolus injection), the approximate tumor mid-line will be imaged during breath holdings until complete tumor enhancement is achieved (approximately 30-40 seconds post injection), followed by imaging sweeps through the tumor. Sweeps will then be acquired in the plane perpendicular to the original, before returning to the original plane. Imaging will be continued until either the onset of contrast washout is observed, or 90 seconds after the contrast injection if no definite contrast washout is observed. The mass will then be intermittently imaged (for 10-15 s) every minute until near complete contrast dissipation is determined (5-7 minutes after contrast injection).

Following a 10 minute Lumason wash-out period, participants will then receive a bolus injection (0.5-1.0 ml) of Sonazoid. Imaging of Sonazoid will be identical to the protocol described above for the first 60 seconds to evaluate arterial phase enhancement. Imaging sweeps (5-10 seconds) of the tumor will then be obtained in at 1 and 2 minutes to evaluate enhancement within the late vascular phase and detect early washout. After that imaging will resume 8-10 minutes after contrast injection to evaluate the Kupffer phase of contrast enhancement. This intermittent imaging scheme is employed to minimize bubble destruction. Of note, contrast agent randomization (Lumason vs. Sonazoid) cannot be achieved in this workflow given the > 2 hour hepatic retention of Sonazoid. Following completion of the exam, patients will be monitored for at least 30 minutes before being discharged and all data will be exported for later off-line analysis. Imaging data will then be used to address the three specific aims.

The research material obtained for this study will include ultrasound images, patient demographics, contrast-enhanced MRI or CT exams, cone beam CT exams during treatment guidance and post-TARE, angiography exams in patients undergoing retreatment, and pathology for patients who go to transplant. Ultrasound studies are being acquired specifically for the purposes of this study, while all other data will be acquired based on the clinical standard of care. All clinical information will be collected by the clinical research coordinators who will maintain the database with individually identifiable private information about human subjects. The information will be maintained on the research coordinators' password protected and encrypted computer. A copy of the database will also be maintained on the principal investigator's computer (secured in the same manner).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for TARE therapy of a treatment naïve HCC visible on ultrasound.
* Be at least 18 years of age.
* Be medically stable.
* If a female of child-bearing age, must have a negative pregnancy test.
* Have signed Informed Consent to participate in the study.

Exclusion Criteria:

* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable.
* Patients with known sensitivities to the components of Lumason.
* Patients with known sensitivities to the components of Sonazoid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor viability on contrast enhanced ultrasound using a blood pooling contrast agent | 1-2 months post treatment
  Viability of tumor assessed by three radiologists using contrast-enhanced ultrasound
Tumor viability on contrast enhanced ultrasound using a blood pooling contrast agent | 3-6 months post treatment
  Viability of tumor assessed by three radiologists using contrast-enhanced ultrasound

SECONDARY OUTCOMES:
Tumor viability on contrast enhanced ultrasound using a Kupffer cell-specific contrast agent | 1-2 months post treatment
  Viability of tumor assessed by three radiologists using contrast-enhanced ultrasound
Tumor viability on contrast enhanced ultrasound using a Kupffer cell-specific contrast agent | 3-6 months post treatment
  Viability of tumor assessed by three radiologists using contrast-enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: John Eisenbrey, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No